CLINICAL TRIAL: NCT06848556
Title: A Multicenter, Randomized, Controlled, Open-label Phase I/II Study to Evaluate the Pharmacokinetics of Transarterial Tirapazamine Embolization for Intermediate-stage Hepatocellular Carcinoma, and Compare Its Efficacy and Safety with Transarterial Chemoembolization
Brief Title: Evaluate the Effect of Tirazamine on Primary Liver Cancer.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Operational Strategy Adjustment
Sponsor: Zhejiang Raygene Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT005
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: TATE; TACE; pharmacokinetics; HEPATOCELLULAR CARCINOMA
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tirapazamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TATE (Experimental): Part one is a multicenter, open-label, dose-escalation clinical trial. The starting dose of Tirapazamine was 5 mg/m² (for 3 patients), followed by 10 mg/m² (for 3 patients) and 20 mg/m² (for 6 patients). All patients received Tirapazamine injected into the hepatic artery that supplies the tumor, followed by an injection of iodized oil, a mixture of gelatin sponge and contrast agent to complete the embolization.
  Part Two is a Phase II open-label, randomized, controlled trial. Patients in the experimental group (Group A) will using a fixed dose of 35 mg of tirapazamine injected into the hepatic artery that supplies the tumor, followed by an injection of iodized oil, a mixture of gelatin sponge and contrast agent to complete the embolization.
  Interventions: Drug: tirapazamine; Procedure: Transarterial Embolization
- TACE (Experimental): Part Two: Patients in the control group (Group B) received standard Transarterial Chemoembolization (TACE) with intra-arterial injection of a mixture of epirubicin and iodized oil at a personalized dose, followed by embolization completed by injecting a suspension of gelatin sponge and contrast agent.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: tirapazamine — Intra-arterial injection into the tumor feeding artery
  Arms: TATE
Procedure: Transarterial Embolization — Lipiodol and Gelfoam used to embolize tumor vessels and induce tumor hypoxia
  Other Names: TAE
  Arms: TATE
Procedure: TACE — Patients received standard Transarterial Chemoembolization (TACE) with intra-arterial injection of a mixture of epirubicin and iodized oil at a personalized dose, followed by embolization completed by injecting a suspension of gelatin sponge and contrast agent.
  Other Names: Transarterial Chemoembolization
  Arms: TACE

SUMMARY:
This Phase I/II trial aims to evaluate the pharmacokinetics, efficacy, and safety of tirapazamine administered via hepatic artery injection followed by TACE in patients with intermediate-stage HCC. The trial will compare the outcomes of TATE with standard TACE.

DETAILED DESCRIPTION:
The clinical trial is bifurcated into two distinct strata.

Phase One:

This stratum is designed to elucidate the pharmacokinetics of Tirapazamine, specifically its concentration in peripheral blood, in patients with hepatocellular carcinoma (HCC) subsequent to hepatic arterial infusion of Tirapazamine at dosages of 5, 10, and 20 mg/m², culminating in hepatic arterial embolization. A total of approximately 12 patients are slated for enrollment, with 3 to 6 patients allocated to each dosage tier. This constitutes a multicenter, open-label, dose-escalation study. Initiation occurs at a Tirapazamine dosage of 5 mg/m² (administered to 3 patients), followed by escalation to 10 mg/m² (administered to 3 patients), and culminating at 20 mg/m² (administered to 6 patients). All subjects undergo hepatic arterial infusion of Tirapazamine directed towards the tumor vasculature, followed by embolization utilizing a formulation comprising iodized oil, gelatin sponge, and contrast agent (the preparation and application of the embolic agent are delineated in Appendix E).

Phase Two:

Phase Two is delineated as a Phase II open-label, randomized, controlled trial that compares the therapeutic outcomes of TATE (Transarterial Tirapazamine Embolization) and TACE (Transarterial Chemoembolization) in patients with intermediate-stage primary hepatocellular carcinoma who are candidates for hepatic arterial embolization. This phase may be conducted contemporaneously with Phase One. Approximately 200 patients will be randomized in a 1:1 ratio to either the experimental arm (Group A, TATE ) or the control arm (Group B, TACE ). Inter-arm crossover is proscribed.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma, either histologically/cytologically confirmed or clinically diagnosed
* Age 18-80 years
* Patient is eligible to do TAE or TACE treatment.
* ECOG performance status score 0-1.
* Child-Pugh score 5 - 7 .
* No portal vein tumor thrombus, lymph node metastasis, peritoneal tumor seeding, or extrahepatic metastasis.

Exclusion Criteria:

* Prior liver transplantation
* History of liver tumor embolization or radioembolization
* Uncontrolled HBV or HCV infection
* Significant cardiovascular, pulmonary, or renal disease
* QTc prolongation or use of QTc-prolonging medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours post-first dose
  Part I: One of the Pharmacokinetic Characteristics
Area under the plasma concentration versus time curve (AUC) | 24 hours post-first dose
  Part I: One of the Pharmacokinetic Characteristics
Time to Maximum Concentration（Tmax） | 24 hours post-first dose
  Part I: One of the Pharmacokinetic Characteristics
Terminal Elimination Half-life（T1/2） | 24 hours post-first dose
  Part I: One of the Pharmacokinetic Characteristics
PFS | 36 months
  Part two:
  Compare the difference in progression-free survival of patients after TATE/TACE treatment to evaluate whether TATE is superior to traditional TACE.

SECONDARY OUTCOMES:
OS | 36 months
  OS defined as the time from randomization to death
CR | 36 months
  The percentage (%) of patients who achieve a complete response (CR) according to the mRECIST criteria after TACE/TATE treatment.
ORR | 36 months
  objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Caifang Ni, M.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Protection of participant privacy